CLINICAL TRIAL: NCT04489277
Title: Silent Brain Infarction After Endovascular Arch Procedures: Preliminary Results From the STEP Registry
Brief Title: Silent Brain Infarction After Endovascular Arch Procedures
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Fondation Hôpital Saint-Joseph (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Vascular Surgical Research Group, Imperial College, London, UK (Unknown); Sanger Heart and Vascular Institute, Charlotte, NC (Unknown); Loyola University Medical Center, Maywood, IL (Unknown); UAB School of Medicine, Birmingham, AL (Unknown); Heidelberg University Hospital, Heidelberg, Germany (Unknown); University Hospital of Freiburg, Freiburg, Germany (Unknown); Stanford University (Other); Massachusetts General Hospital (Other); Baylor Research Hospital, Dallas, TX (Unknown); Emory University Hospital, Atlanta, GA (Unknown); University Hospital of Mainz, Mainz, Germany (Unknown); Diakonie Hospital Jung-Stilling, Siegen, Germany (Unknown); Mayo Clinic, Rochester, MN (Unknown); Sentara Vascular/Eastern Virginia Medical School, Norfolk, VA (Unknown); Maastricht University Medical Centre, Maastricht, Netherlands (Unknown); I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Italy (Unknown); Memorial Care Long Beach Heart & Vascular Institute, Long Beach, CA (Unknown)
Responsible Party: Principal Investigator, Wolf Eilenberg, Professor Stephan Haulon, Proessor Tilo Kölbel, Fondation Hôpital Saint-Joseph
Other Study IDs: INSERM UMR_S 999
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Aortic Arch Aneurysm
Keywords: Thoracic endovascular aortic repair; Silent cerebral infarction; Stroke; Magnetic resonance imaging; DW-MRI; Aortic arch disease
MeSH Terms: conditions — Aneurysm, Aortic Arch; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 17 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Silent Brain Infarction: treated with an aortic endoprosthesis deployed in Ishimaru zone 0 to 3 and brain diffusion-weighted magnetic resonance imaging (DW-MRI) within 7 days after the procedure with silent brain infarction
  Interventions: Device: Endovascular Arch Procedures
- Patients without Silent Brain Infarction: treated with an aortic endoprosthesis deployed in Ishimaru zone 0 to 3 and brain diffusion-weighted magnetic resonance imaging (DW-MRI) within 7 days after the procedure without silent brain infarction
  Interventions: Device: Endovascular Arch Procedures

INTERVENTIONS:
Device: Endovascular Arch Procedures — Endovascular Arch Procedures (TEVAR, Branch endografts, Fenestrated endografts)

SUMMARY:
This is the largest study to evaluate incidence and distribution of silent cerebral infarction (SBI) following endovascular repair for disease of the aortic arch. Also, it is the first cohort to include total endovascular arch repair and devices flushed with carbon dioxide (CO2) to prevent gaseous cerebral embolization.

DETAILED DESCRIPTION:
Introduction. Poor data exist concerning the rate of silent cerebral ischemic events following endovascular treatment of the aortic arch. The objective of this work was to quantify these lesions using the STEP registry.

Methods. This multicentre retrospective cohort study included consecutive patients treated with an aortic endoprosthesis deployed in Ishimaru zone 0 to 3 and brain diffusion-weighted magnetic resonance imaging (DW-MRI) within 7 days after the procedure. DW-MRI was performed to identify the location and number of new silent brain infarctions (SBI), microbleeds ans general outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Included patients underwent a proximal endograft deployment in Ishimaru zone 0 to 3

Exclusion Criteria:

* Missing preoperative computed tomography angiography (CTA) scan of the chest and any circumstances that precluded the DW-MRI to be performed in the appropriate time window, such as a medical condition or an MRI contraindication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients, who received routine postoperative DW-MRI within 7 days after endovascular aortic arch repair between September 2018 and January 2020 at the University Hospital Hamburg-Eppendorf (Hamburg, Germany) and Marie Lannelongue Hospital (Paris, France) were identified.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
frequency of silent cerebral infarcts on DW-MRI | 7 days
  Primary outcomes were the frequency of silent cerebral infarcts on DW-MRI after endovascular arch procedures, and to identify the number, the distribution, and predictors of these lesions.

SECONDARY OUTCOMES:
perioperative ischemic stroke | 30 days
  Secondary outcomes were perioperative ischemic stroke defined as a brain infarction of ischemic etiology which occurs during surgery or within 30 days after surgery, TIA, hemorrhagic stroke, 30-day mortality, spinal cord ischemia, length of stay and discharge disposition.

CONTACTS AND LOCATIONS:
Locations (2):
- Marie Lannelongue Hospital (Paris, France), Paris, France
- University Hospital Hamburg-Eppendorf (Hamburg, Germany), Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charbonneau P, Kolbel T, Rohlffs F, Eilenberg W, Planche O, Bechstein M, Ristl R, Greenhalgh R, Haulon S; STEP collaborators. Silent Brain Infarction After Endovascular Arch Procedures: Preliminary Results from the STEP Registry. Eur J Vasc Endovasc Surg. 2021 Feb;61(2):239-245. doi: 10.1016/j.ejvs.2020.11.021. Epub 2020 Dec 22. PMID 33358103